CLINICAL TRIAL: NCT03346096
Title: TEAM (Thiotepa, Etoposide, Cytosar, Melphalan ) in Preparation for Autologous Hematopoietic Stem-Cell Transplantation in Patients With Non-Hodgkin's and Hodgkin's Lymphoma.
Brief Title: TEAM (Thiotepa, Etoposide, Cytosar, Melphalan ) for AutoSCT in Lymphoma
Acronym: TEAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sheba - 17 - 4053 - AN - CTIL
Record Dates: First submitted 2017-10-15; First posted 2017-11-17 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Malignant Lymphoma
Keywords: TEAM (Thiotepa, Etoposide, Cytosar, Melphalan ); autologous stem-cell transplantation (ASCT); malignant lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Thiotepa

STUDY DESIGN:
Intervention Model Description: TEAM conditioning consisted of THIOTEPA 5mg/kg on days -7-6, etoposide 200 mg/m2 , Cytosar (ARA-C) 200 mg/m2 on days -5,-4, -3, -2 and melphalan 140 mg/m2 on day -1 followed by autologous hematopoietic stem-cell transplantation as per standard institutional protocols.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thiotepa (Experimental): Thiotepa for reduce toxicity and improve outcome following transplantation
  Interventions: Drug: Thiotepa

INTERVENTIONS:
Drug: Thiotepa — fixed dose 5mg/kg on days -7-6

SUMMARY:
Study is designed to explore whether the introduction of Thiotepa, to the pre autologous stem-cell transplantation (ASCT) conditioning will reduce toxicity and thus improve outcome following transplantation in up to 24 patients with malignant lymphoma including both non-Hodgkin's lymphoma (NHL) and Hodgkin's lymphoma ( HL) improving toxicity profile , reducing side effects while potentially improving the antitumor response. Specifically,we speculate that using the novel Thiotepa based TEAM consisted of THIOTEPA 5mg/kg on days -7-6, etoposide 200 mg/m2 , Cytosar (ARA-C) 200 mg/m2 on days -5,-4, -3, -2 and melphalan 140 mg/m2 on day -1, pre transplantation conditioning regimen may allow transplantation with lower transplant related toxicity and thus improve outcome in this setting. Toward this aim the impact on toxicity profile ,engraftment and disease control will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-Hodgkin's and Hodgkin's lymphoma as confirmed by a pathological biopsy report.
2. Patients who are candidates for Autologous stem-cell transplantation due to refractory or relapsing disease by standard institutional indications and comply with standard transplant eligibility criteria.
3. Age less than physiologic 70 years.
4. Patients with an adequate autologous stem cell collection for transplantation and backup (>5 x 106 CD34(cluster of differentiation 34)+ cells/kg) .Patients must sign written informed consent.
5. No limitation on bulky disease or bone marrow involvement. No limitation on the number and response to prior therapy. Prior autologous transplantation and/or treatment with rituximab allowed. All prior chemotherapy completed at least three weeks before study treatment

Exclusion Criteria:

1. Bilirubin > 3.0 mg/dl, transaminases > 3 times upper normal limit
2. Creatinine > 2.0 mg/dl
3. Eastern Cooperative Oncology Group (ECOG) Performance status > 2
4. Uncontrolled infection
5. Pregnancy or lactation
6. Abnormal lung diffusion capacity (DLCO < 40% predicted)
7. Severe cardiovascular disease
8. CNS (central nervous system) disease involvement
9. Pleural effusion or ascites > 1 liter
10. Psychiatric conditions/disease that impair the ability to give informed consent or to adequately co-operate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Toxicities graded by Bearman's criteria and infectious complications | 15 month
  To determine the relative toxicity and response rate of TEAM preparative regimen pre- Autologous stem cell transplantation in patients with non-Hodgkin's and Hodgkin's Lymphoma

CONTACTS AND LOCATIONS:
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel